CLINICAL TRIAL: NCT00596037
Title: A Phase III, Open-label, Uncontrolled, Multicentre, Rollover Study to Assess Safety and Efficacy of LB03002 Administered Weekly in Adults With Growth Hormone Deficiency
Brief Title: Treatment of Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Collaborators: BioPartners GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPLG-005-RO
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Pituitary Disorders; Adult Growth Hormone Deficiency
Keywords: Growth hormone Deficiency
MeSH Terms: conditions — Pituitary Diseases; Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LB03002 throughout (Experimental): administered LB03002 for preceding 26 weeks
  Interventions: Drug: Growth hormone - LB03002
- Switched to LB03002 (Experimental): administered placebo for preceding 26 weeks
  Interventions: Drug: Growth hormone - LB03002

INTERVENTIONS:
Drug: Growth hormone - LB03002

SUMMARY:
The objective of this rollover study is to evaluate the long term (1 year) safety of a new weekly administered growth hormone preparation in adults with growth hormone deficiency who were treated with the same experimental preparation in study BPLG-005. In addition, further change in efficacy endpoints of BPLG-005 by prolonged treatment will be evaluated. Additional efficacy and safety data of the experimental preparation will be obtained from the switch-over patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) who have completed the Visit 8 of preceding main study (BPLG-005) and are willing to continue their participation in an extension study
* If female, women of child-bearing potential who are using a reliable method of contraception and be willing to use it throughout the study. A negative urine pregnancy test at Visit 0 is required for females of child-bearing potential
* Written informed consent of the patient

Exclusion Criteria:

* Evidence of active malignancy or growth of a previously stable tumor
* Benign intracranial hypertension
* Clinically significant respiratory, cardiac, hepatic, renal, neuromuscular disease
* Non-compliance with medications, un-cooperativeness or drug abuse during the BPLG-005 study
* Patients who are not able to comply with the study protocol for any reason

Ages: 23 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, antibody formation and local tolerability assessment after 1 year treatment from baseline of BPLG-005 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: HJ Ji, PhD, Study Chair — LG Life Sciences